CLINICAL TRIAL: NCT01451502
Title: Infusion of Cell Populations From Unlicensed Umbilical Cord Blood Units
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011LS079; MT2011-13R (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2011-10-11; First posted 2011-10-13 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Lymphatic Diseases; Hematopoietic Malignancy
Keywords: umbilical cord blood
MeSH Terms: conditions — Lymphatic Diseases; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Unlicensed Umbilical Cord Blood Infusion (Experimental): All patients will be registered in OnCore under this protocol as well as the specific treatment protocol.
  * Pre-infusion treatment using intravenous hydration, acetaminophen and diphenhydramine hydrochloride
  * Unlicensed Umbilical Cord Blood Infusion according to institutional guidelines.
    * Infusion of minimally manipulated unlicensed UCB units:
    * vital signs Monitoring during and after UCB infusion:
    * Management of infusion reactions
  * Post-transplant care and follow-up: will be done according to the disease specific treatment protocol and institutional guidelines.
  Interventions: Biological: Umbilical Cord Blood (UCB)

INTERVENTIONS:
Biological: Umbilical Cord Blood (UCB) — Infusion of Minimally Manipulated UCB Units - the UCB unit will be infused through a central line according to institutional guidelines.

SUMMARY:
For the next 5-10 years or possibly longer, a high proportion of the Cord Blood Banks (CBB) inventory worldwide will be composed of unlicensed umbilical cord blood (UCB) units. While Food and Drug Administration (FDA)-licensed units will be prioritized, it will always be possible that an unlicensed unit will have known attributes, making it a better source of cells for the given indication. Because of the wide variety of current and potential indications as a source of cells for hematopoietic reconstitution or other form of cellular therapy, it is critical that the investigators have access to unlicensed UCB units.

DETAILED DESCRIPTION:
Patients will receive intravenous hydration, acetaminophen and diphenhydramine hydrochloride (or appropriate alternative regimen) approximately 30 minutes prior to UCB infusion with doses adjusted for subject age and weight unless otherwise specified in the specific treatment protocol. Additional treatments will vary with the specific use of the UCB cells as specified in institutional review board (IRB)-approved disease-specific protocols at the University of Minnesota.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for an unlicensed umbilical cord blood (UCB) unit, the subject must meet each of the eligibility criteria listed below:

* Subjects with any diagnosis for which there is an institutional review board (IRB) approved treatment protocol that requires UCB as a source of hematopoietic stem cells for lympho-hematopoietic reconstitution after myeloablative or non myeloablative conditioning.
* Subject (or parent/guardian) must provide written informed consent for the use of unlicensed UCB units with co-enrollment onto a University of Minnesota IRB-approved clinical trial that details the disease specific treatment plan that prescribes the use of UCB as source of cells
* Subject has an unlicensed UCB unit that meets required cell dose and HLA matching criteria (as defined in the primary treatment protocol) that is considered negative for tested blood-borne pathogens and also lack an 'equivalent', licensed UCB unit from a University of Minnesota approved Cord Blood Bank

Exclusion Criteria:

* Exclusion criteria are specified in the treatment protocol according to indication.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2011-10-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Blood Borne Pathogen Transmission from Unlicensed UCB Units. | Within 24 Hours Post Infusion
  Documentation of events for the purpose of this study will only be for those events at least possibly related to the unlicensed UCB. Monitoring for acute infusional toxicities will end 24 hours after the umbilical cord blood (UCB) infusion.

SECONDARY OUTCOMES:
Incidence of Serious Infusion Reactions of Minimally Manipulated Unlicensed UCB Units | Up to Day 180
  point estimations and 95% confidence intervals of serious infusion reaction
Number of the Desired Lineage Specific Cells in Minimally Manipulated Unlicensed UCB Units | Prior to Infusion
  Upon thawing (e.g., number of CD34 and colony forming cells for hematopoietic products or number of CD4+/CD25+/CD127- cells for Treg products prior to further manipulation).
Incidence of Mislabeled UCB Units | Up to Day 180
  Point estimations and 95% confidence intervals of incidences mislabeled UCB units
Comparison of Specific Cord Blood Banks (CBBs) | Up to Day 180
  Determine if bacterial contamination, poor cell recoveries, shipment of mislabeled units, blood borne pathogen transmission or serious infusion reactions are more prevalent in units from specific CBBs.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Hoover, MD, MSc, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States